CLINICAL TRIAL: NCT00831844
Title: A Phase II Study of IMC-A12 (Anti-IGF-I Receptor Monoclonal Antibody, NSC #742460) in Children With Relapsed/Refractory Solid Tumors
Brief Title: Cixutumumab in Treating Patients With Relapsed or Refractory Solid Tumors
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-01170; NCI-2009-01170 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000633186 (Other: Clinical Trials.gov); COG-ADVL0821 (Other: Children's Oncology Group); ADVL0821 (Other: Children's Oncology Group); ADVL0821 (Other: CTEP); U10CA098543 (NIH)
Record Dates: First submitted 2009-01-28; First posted 2009-01-29 (Estimated); Results first posted 2015-03-30 (Estimated); Last update posted 2015-03-30 (Estimated); Status verified 2015-03

CONDITIONS: Adult Rhabdomyosarcoma; Adult Synovial Sarcoma; Childhood Hepatoblastoma; Childhood Synovial Sarcoma; Previously Treated Childhood Rhabdomyosarcoma; Recurrent Adrenocortical Carcinoma; Recurrent Adult Soft Tissue Sarcoma; Recurrent Childhood Liver Cancer; Recurrent Childhood Rhabdomyosarcoma; Recurrent Childhood Soft Tissue Sarcoma; Recurrent Ewing Sarcoma/Peripheral Primitive; Neuroectodermal Tumor; Recurrent Neuroblastoma; Recurrent Osteosarcoma; Recurrent Retinoblastoma; Recurrent Wilms Tumor and Other Childhood Kidney Tumors
MeSH Terms: conditions — Rhabdomyosarcoma; Sarcoma, Synovial; Hepatoblastoma; Adrenocortical Carcinoma; Sarcoma; Sarcoma, Ewing; Neuroectodermal Tumors; Neuroblastoma; Osteosarcoma; Retinoblastoma; Wilms Tumor | interventions — cixutumumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (10):
- Group 1 - Recurrent or Refractory Hepatoblastoma (Experimental): Group 1 - Recurrent or Refractory Hepatoblastoma. Patients receive cixutumumab IV over 1 hour on days 1, 8, 15, and 22. Treatment repeats every 28 days for up to 24 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: cixutumumab; Other: laboratory biomarker analysis
- Group 2 - Recurrent or Refractory Synovial Sarcoma (Experimental): Group 2 - Recurrent or Refractory Synovial Sarcoma. Patients receive cixutumumab IV over 1 hour on days 1, 8, 15, and 22. Treatment repeats every 28 days for up to 24 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: cixutumumab; Other: laboratory biomarker analysis
- Group 3 - Recurrent or Refractory Rhabdomyosarcoma (Experimental): Group 3 - Recurrent or Refractory Rhabdomyosarcoma. Patients receive cixutumumab IV over 1 hour on days 1, 8, 15, and 22. Treatment repeats every 28 days for up to 24 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: cixutumumab; Other: laboratory biomarker analysis
- Grp 4-Recurrent or Refractory Adrenocortical Carcinoma (Experimental): Group 4 - Recurrent or Refractory Adrenocortical Carcinoma. Patients receive cixutumumab IV over 1 hour on days 1, 8, 15, and 22. Treatment repeats every 28 days for up to 24 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: cixutumumab; Other: laboratory biomarker analysis
- Grp 5-Ewing Sarcoma/Peripheral Primitive Neuroectodermal Tumor (Experimental): Group 5 - Recurrent or Refractory Ewing Sarcoma/Peripheral Primitive Neuroectodermal Tumor. Patients receive cixutumumab IV over 1 hour on days 1, 8, 15, and 22. Treatment repeats every 28 days for up to 24 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: cixutumumab; Other: laboratory biomarker analysis
- Grp 6 - Neuroblastoma-MIBG Positive Without Measurable Disease (Experimental): Group 6 - Recurrent or Refractory Neuroblastoma -meta-iodobenzylguanidine (MIBG) Positive Without Measurable Disease. Patients receive cixutumumab IV over 1 hour on days 1, 8, 15, and 22. Treatment repeats every 28 days for up to 24 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: cixutumumab; Other: laboratory biomarker analysis
- Grp 7-Neuroblastoma with measurable disease (Experimental): Group 7 - Recurrent or Refractory Neuroblastoma -With Measurable Disease. Patients receive cixutumumab IV over 1 hour on days 1, 8, 15, and 22. Treatment repeats every 28 days for up to 24 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: cixutumumab; Other: laboratory biomarker analysis
- Group 8 - Recurrent Osteosarcoma (Experimental): Group 8 - Recurrent Osteosarcoma. Patients receive cixutumumab IV over 1 hour on days 1, 8, 15, and 22. Treatment repeats every 28 days for up to 24 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: cixutumumab; Other: laboratory biomarker analysis
- Group 9 - Recurrent or Refractory Wilms Tumor (Experimental): Group 9 - Recurrent or Refractory Wilms Tumor. Patients receive cixutumumab IV over 1 hour on days 1, 8, 15, and 22. Treatment repeats every 28 days for up to 24 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: cixutumumab; Other: laboratory biomarker analysis
- Group 10 - Recurrent or Refractory Retinoblastoma (Experimental): Group 10 - Recurrent or Refractory Retinoblastoma. Patients receive cixutumumab IV over 1 hour on days 1, 8, 15, and 22. Treatment repeats every 28 days for up to 24 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: cixutumumab; Other: laboratory biomarker analysis

INTERVENTIONS:
Biological: cixutumumab — Given IV: Week 1 day 1, 9 mg/kg/dose over 1 hour. Week 2 Day 8, 9 mg/kg/dose over 1 hour. Week 3 Day 15, 9 mg/kg/dose over 1 hour. Week 4 Day 22, 9 mg/kg/dose over 1 hour.
  Other Names: anti-IGF-1R recombinant monoclonal antibody IMC-A12; IMC-A12
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This phase II trial is studying the side effects and how well cixutumumab works in treating patients with relapsed or refractory solid tumors. Monoclonal antibodies, such as cixutumumab, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the response rate to IMC-A12 (cixutumumab) administered in various strata of recurrent/refractory malignant solid tumors in childhood and young adulthood.

II. To further define and describe the toxicities of IMC-A12. III. To further characterize the pharmacokinetics of IMC-A12.

SECONDARY OBJECTIVES:

I. To examine the relationship between tumor expression of insulin-like growth factor (IGF)-I, IGF-II, and IGF-I receptor (IR) and response to IMC-A12.

II. To determine the human anti-human antibody (HAHA) response after treatment with IMC-A12.

III. To further evaluate the effect of IMC-A12 on circulating levels of proteins involved in linear growth and glucose homeostasis, including IGF-I, IGF-II, IGF-BP3, growth hormone, insulin, and C-peptide.

OUTLINE: This is a multicenter study. Patients are stratified according to disease type.

Patients receive cixutumumab intravenously (IV) over 1 hour on days 1, 8, 15, and 22. Treatment repeats every 28 days for up to 24 courses in the absence of disease progression or unacceptable toxicity.

Patients undergo blood sample collection periodically for correlative laboratory studies. Samples are analyzed for IGF-I, IGF-II, IGF-BP3, growth hormone, insulin, and C-peptide levels and for immunogenicity.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed malignant solid tumor, including the following:

  * Osteosarcoma
  * Ewing sarcoma/peripheral primitive neuroectodermal tumor
  * Rhabdomyosarcoma
  * Neuroblastoma
  * Wilms tumor
  * Synovial sarcoma
  * Hepatoblastoma
  * Adrenocortical carcinoma
  * Retinoblastoma
* No known curative therapy or therapy proven to prolong survival with an acceptable quality of life exists
* Radiographically measurable disease*, defined as ≥ 1 unidimensionally measurable lesion ≥ 20 mm by MRI or CT scan or ≥ 10 mm by spiral CT scan

  * The following are not considered measurable disease:

    * Ascites, pleural effusions, or other malignant fluid collections
    * Bone marrow infiltration by tumor
    * Lesions detected only by non-MIBG nuclear medicine studies (e.g., bone scan)
    * Previously irradiated lesions that have not demonstrated clear progression post-radiotherapy
* No known Central Nervous System (CNS) metastases unless they were treated by surgery or radiotherapy AND are stable with no recurrent lesions for ≥ 3 months
* Lansky or Karnofsky performance status (PS) 50-100% OR Eastern Cooperative Oncology Group (ECOG) PS 0-2
* Absolute neutrophil count (ANC) ≥ 1,000/mm³ (> 250/mm³ for patients with neuroblastoma)
* Platelet count ≥ 75,000/mm³ (> 25,000/mm³ for patients with neuroblastoma) (transfusion independent)
* Hemoglobin ≥ 8.0 g/dL (≥ 7.5 g/dL for patients with neuroblastoma) (RBC transfusion allowed)
* Creatinine clearance or radioisotope glomerular filtration rate ≥ 70 mL/min OR serum creatinine normal based on age/gender as follows:

  * ≤ 0.4 mg/dL (for patients 1 to 5 months of age)
  * ≤ 0.5 mg/dL (for patients 6 to 11 months of age)
  * ≤ 0.6 mg/dL (for patients 1 year of age)
  * ≤ 0.8 mg/dL (for patients 2 to 5 years of age)
  * ≤ 1 mg/dL (for patients 6 to 9 years of age)
  * ≤ 1.2 mg/dL (for patients 10 to 12 years of age)
  * ≤ 1.5 mg/dL (males) or 1.4 mg/dL (females) (for patients 13 to 15 years of age)
  * ≤ 1.7 mg/dL (males) or 1.4 mg/dL (females) (for patients ≥ 16 years of age)
* Total bilirubin ≤ 1.5 times upper limit of normal for age
* Alanine transaminase (ALT) ≤ 110 U/L
* Serum albumin ≥ 2 g/dL
* Blood glucose normal
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 3 months after completion of study treatment
* Able to comply with safety monitoring requirements of study
* No history of allergic reactions attributed to compounds of similar chemical or biologic composition to study drug
* No uncontrolled infection
* No known type I or II diabetes mellitus
* Recovered from prior chemotherapy, immunotherapy, or radiotherapy
* More than 3 weeks since prior myelosuppressive chemotherapy (6 weeks for nitrosoureas)
* At least 7 days since prior hematopoietic growth factors (14 days for pegfilgrastim)
* At least 6 weeks since prior monoclonal antibody therapy
* At least 7 days since other prior antineoplastic biologic agents
* No prior monoclonal antibody targeting the IGF-IR
* No prior small molecule kinase inhibitors of IGF-IR
* At least 2 weeks since prior local palliative (small port) radiotherapy
* At least 3 months since prior total-body irradiation, craniospinal radiotherapy, or radiotherapy to ≥ 50% of the pelvis
* At least 6 weeks since other prior substantial bone marrow radiotherapy
* At least 2 months since prior stem cell transplantation

  * No evidence of graft-versus-host disease
* Concurrent corticosteroids allowed provided dose is stable or decreasing over the past 7 days

  * Intermittent use of corticosteroids to manage infusional reactions allowed
* No other concurrent anticancer therapy, including chemotherapy, radiotherapy, immunotherapy, or biologic therapy
* No other concurrent investigational agents
* No concurrent insulin or growth hormone therapy

Ages: 7 Months to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 116 (Actual)
Dates: Start 2009-01; Primary Completion 2013-04 (Actual); Study Completion 2013-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brenda Weigel, MD, Principal Investigator — Children's Oncology Group
Locations (105):
- United States (93):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Southern California Permanente Medical Group, Downey, California
  - Miller Children's Hospital, Long Beach, California
  - Children's Hospital Los Angeles, Los Angeles, California
  - Children's Hospital Central California, Madera, California
  - Kaiser Permanente-Oakland, Oakland, California
  - Childrens Hospital of Orange County, Orange, California
  - Lucile Packard Children's Hospital Stanford University, Palo Alto, California
  - University of California San Francisco Medical Center-Parnassus, San Francisco, California
  - Connecticut Children's Medical Center, Hartford, Connecticut
  - Alfred I duPont Hospital for Children, Wilmington, Delaware
  - Lombardi Comprehensive Cancer Center at Georgetown University, Washington D.C., District of Columbia
  - Lee Memorial Health System, Fort Myers, Florida
  - Nemours Children's Clinic - Jacksonville, Jacksonville, Florida
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - Miami Children's Hospital, Miami, Florida
  - Florida Hospital, Orlando, Florida
  - Nemours Childrens Clinic - Orlando, Orlando, Florida
  - UF Cancer Center at Orlando Health, Orlando, Florida
  - Nemours Children's Clinic - Pensacola, Pensacola, Florida
  - All Children's Hospital, St. Petersburg, Florida
  - Saint Joseph Children's Hospital of Tampa, Tampa, Florida
  - Saint Mary's Hospital, West Palm Beach, Florida
  - Children's Healthcare of Atlanta - Egleston, Atlanta, Georgia
  - University of Hawaii, Honolulu, Hawaii
  - Saint Luke's Mountain States Tumor Institute, Boise, Idaho
  - University of Illinois, Chicago, Illinois
  - Lurie Children's Hospital-Chicago, Chicago, Illinois
  - University of Chicago, Chicago, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Saint Jude Midwest Affiliate, Peoria, Illinois
  - Southern Illinois University, Springfield, Illinois
  - Indiana University Medical Center, Indianapolis, Indiana
  - University of Kentucky, Lexington, Kentucky
  - Sinai Hospital of Baltimore, Baltimore, Maryland
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - C S Mott Children's Hospital, Ann Arbor, Michigan
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Saint John Hospital and Medical Center, Detroit, Michigan
  - Helen DeVos Children's Hospital at Spectrum Health, Grand Rapids, Michigan
  - Children's Hospitals and Clinics of Minnesota - Minneapolis, Minneapolis, Minnesota
  - University of Minnesota Medical Center-Fairview, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - University of Missouri - Ellis Fischel, Columbia, Missouri
  - The Childrens Mercy Hospital, Kansas City, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Children's Hospital and Medical Center of Omaha, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Nevada Cancer Research Foundation CCOP, Las Vegas, Nevada
  - Hackensack University Medical Center, Hackensack, New Jersey
  - UMDNJ - Robert Wood Johnson University Hospital, New Brunswick, New Jersey
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Albany Medical Center, Albany, New York
  - New York University Langone Medical Center, New York, New York
  - Columbia University Medical Center, New York, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - University of Rochester, Rochester, New York
  - State University of New York Upstate Medical University, Syracuse, New York
  - New York Medical College, Valhalla, New York
  - Carolinas Medical Center, Charlotte, North Carolina
  - Children's Hospital Medical Center of Akron, Akron, Ohio
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Rainbow Babies and Childrens Hospital, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Oregon Health and Science University, Portland, Oregon
  - Lehigh Valley Hospital - Muhlenberg, Bethlehem, Pennsylvania
  - Penn State Hershey Children's Hospital, Hershey, Pennsylvania
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - Palmetto Health Richland, Columbia, South Carolina
  - Greenville Cancer Treatment Center, Greenville, South Carolina
  - T C Thompson Children's Hospital, Chattanooga, Tennessee
  - East Tennessee Childrens Hospital, Knoxville, Tennessee
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee
  - Texas Tech University Health Science Center-Amarillo, Amarillo, Texas
  - Medical City Dallas Hospital, Dallas, Texas
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Cook Children's Medical Center, Fort Worth, Texas
  - Baylor College of Medicine, Houston, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Scott and White Memorial Hospital, Temple, Texas
  - Primary Children's Hospital, Salt Lake City, Utah
  - Childrens Hospital-King's Daughters, Norfolk, Virginia
  - Virginia Commonwealth University, Richmond, Virginia
  - Seattle Children's Hospital, Seattle, Washington
  - Providence Sacred Heart Medical Center and Children's Hospital, Spokane, Washington
  - Mary Bridge Children's Hospital and Health Center, Tacoma, Washington
  - Midwest Children's Cancer Center, Milwaukee, Wisconsin
- Australia (4):
  - The Children's Hospital at Westmead, Westmead, New South Wales
  - Royal Brisbane and Women's Hospital, Herston, Queensland
  - Royal Children's Hospital, Parkville, Victoria
  - Princess Margaret Hospital for Children, Perth, Western Australia
- Canada (8):
  - British Columbia Children's Hospital, Vancouver, British Columbia
  - CancerCare Manitoba, Winnipeg, Manitoba
  - Janeway Child Health Centre, St. John's, Newfoundland and Labrador
  - IWK Health Centre, Halifax, Nova Scotia
  - Hospital for Sick Children, Toronto, Ontario
  - Centre Hospitalier Universitaire Sainte-Justine, Montreal, Quebec
  - Allan Blair Cancer Centre, Regina, Saskatchewan
  - Saskatoon Cancer Centre, Saskatoon, Saskatchewan

RESULTS

PARTICIPANT FLOW:
Recruitment Details: No patients were enrolled in Group 10, recurrent or refractory retinoblastoma.
Groups:
- Group 1 - Recurrent or Refractory Hepatoblastoma: Group 1 - Recurrent or Refractory Hepatoblastoma. Patients receive cixutumumab IV over 1 hour on days 1, 8, 15, and 22. Treatment repeats every 28 days for up to 24 courses in the absence of disease progression or unacceptable toxicity.
  cixutumumab: Given IV
  laboratory biomarker analysis: Correlative studies
- Group 2 - Recurrent or Refractory Synovial Sarcoma: Group 2 - Recurrent or Refractory Synovial Sarcoma. Patients receive cixutumumab IV over 1 hour on days 1, 8, 15, and 22. Treatment repeats every 28 days for up to 24 courses in the absence of disease progression or unacceptable toxicity.
  cixutumumab: Given IV
  laboratory biomarker analysis: Correlative studies
- Group 3 - Recurrent or Refractory Rhabdomyosarcoma: Group 3 - Recurrent or Refractory Rhabdomyosarcoma. Patients receive cixutumumab IV over 1 hour on days 1, 8, 15, and 22. Treatment repeats every 28 days for up to 24 courses in the absence of disease progression or unacceptable toxicity.
  cixutumumab: Given IV
  laboratory biomarker analysis: Correlative studies
- Grp 4-Recurrent or Refractory Adrenocortical Carcinoma: Group 4 - Recurrent or Refractory Adrenocortical Carcinoma. Patients receive cixutumumab IV over 1 hour on days 1, 8, 15, and 22. Treatment repeats every 28 days for up to 24 courses in the absence of disease progression or unacceptable toxicity.
  cixutumumab: Given IV
  laboratory biomarker analysis: Correlative studies
- Grp 5-Ewing Sarcoma/Peripheral Primitive Neuroectodermal Tumor: Group 5 - Recurrent or Refractory Ewing Sarcoma/Peripheral Primitive Neuroectodermal Tumor. Patients receive cixutumumab IV over 1 hour on days 1, 8, 15, and 22. Treatment repeats every 28 days for up to 24 courses in the absence of disease progression or unacceptable toxicity.
  cixutumumab: Given IV
  laboratory biomarker analysis: Correlative studies
- Grp 6 - Neuroblastoma-MIBG Positive Without Measurable Disease: Group 6 - Recurrent or Refractory Neuroblastoma -meta-iodobenzylguanidine (MIBG) Positive Without Measurable Disease. Patients receive cixutumumab IV over 1 hour on days 1, 8, 15, and 22. Treatment repeats every 28 days for up to 24 courses in the absence of disease progression or unacceptable toxicity.
  cixutumumab: Given IV
  laboratory biomarker analysis: Correlative studies
- Grp 7-Neuroblastoma With Measurable Disease: Group 7 - Recurrent or Refractory Neuroblastoma -With Measurable Disease. Patients receive cixutumumab IV over 1 hour on days 1, 8, 15, and 22. Treatment repeats every 28 days for up to 24 courses in the absence of disease progression or unacceptable toxicity.
  cixutumumab: Given IV
  laboratory biomarker analysis: Correlative studies
- Group 8 - Recurrent Osteosarcoma: Group 8 - Recurrent Osteosarcoma. Patients receive cixutumumab IV over 1 hour on days 1, 8, 15, and 22. Treatment repeats every 28 days for up to 24 courses in the absence of disease progression or unacceptable toxicity.
  cixutumumab: Given IV
  laboratory biomarker analysis: Correlative studies
- Group 9 - Recurrent or Refractory Wilms Tumor: Group 9 - Recurrent or Refractory Wilms Tumor. Patients receive cixutumumab IV over 1 hour on days 1, 8, 15, and 22. Treatment repeats every 28 days for up to 24 courses in the absence of disease progression or unacceptable toxicity.
  cixutumumab: Given IV
  laboratory biomarker analysis: Correlative studies
- Group 10 - Recurrent or Refractory Retinoblastoma: Group 10 - Recurrent or Refractory Retinoblastoma. Patients receive cixutumumab IV over 1 hour on days 1, 8, 15, and 22. Treatment repeats every 28 days for up to 24 courses in the absence of disease progression or unacceptable toxicity.
  cixutumumab: Given IV
  laboratory biomarker analysis: Correlative studies
Period: Overall Study
Arm/Group | Group 1 - Recurrent or Refractory Hepatoblastoma | Group 2 - Recurrent or Refractory Synovial Sarcoma | Group 3 - Recurrent or Refractory Rhabdomyosarcoma | Grp 4-Recurrent or Refractory Adrenocortical Carcinoma | Grp 5-Ewing Sarcoma/Peripheral Primitive Neuroectodermal Tumor | Grp 6 - Neuroblastoma-MIBG Positive Without Measurable Disease | Grp 7-Neuroblastoma With Measurable Disease | Group 8 - Recurrent Osteosarcoma | Group 9 - Recurrent or Refractory Wilms Tumor | Group 10 - Recurrent or Refractory Retinoblastoma
Started | 10 | 12 | 21 | 10 | 14 | 20 | 10 | 10 | 9 | 0
Completed | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not Completed | 10 | 12 | 20 | 10 | 14 | 19 | 10 | 10 | 9 | 0
Not completed — Adverse Event | 2 | 0 | 0 | 0 | 1 | 1 | 2 | 0 | 0 | 0
Not completed — Death | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lack of Efficacy | 8 | 10 | 15 | 8 | 11 | 17 | 8 | 9 | 7 | 0
Not completed — Physician Decision | 0 | 1 | 3 | 1 | 1 | 1 | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Not completed — Ineligible | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Group 10, Recurrent or Refractory Retinoblastoma no patients were enrolled.
Groups:
- Grp 6 - Neuroblastoma-MIBG Positive Without Measurable Disease: Group 6 - Recurrent or Refractory Neuroblastoma -MIBG Positive Without Measurable Disease. Patients receive cixutumumab IV over 1 hour on days 1, 8, 15, and 22. Treatment repeats every 28 days for up to 24 courses in the absence of disease progression or unacceptable toxicity.
  cixutumumab: Given IV
  laboratory biomarker analysis: Correlative studies
- Total: Total of all reporting groups
Arm/Group | Group 1 - Recurrent or Refractory Hepatoblastoma | Group 2 - Recurrent or Refractory Synovial Sarcoma | Group 3 - Recurrent or Refractory Rhabdomyosarcoma | Grp 4-Recurrent or Refractory Adrenocortical Carcinoma | Grp 5-Ewing Sarcoma/Peripheral Primitive Neuroectodermal Tumor | Grp 6 - Neuroblastoma-MIBG Positive Without Measurable Disease | Grp 7-Neuroblastoma With Measurable Disease | Group 8 - Recurrent Osteosarcoma | Group 9 - Recurrent or Refractory Wilms Tumor | Group 10 - Recurrent or Refractory Retinoblastoma | Total
Number analyzed (Participants) | 10 | 12 | 21 | 10 | 14 | 20 | 10 | 10 | 9 | 0 | 116
Age, Categorical [Number; unit: participants]
  <=18 years | 10 | 8 | 16 | 8 | 9 | 18 | 7 | 8 | 9 |  | 93
  Between 18 and 65 years | 0 | 4 | 5 | 2 | 5 | 2 | 3 | 2 | 0 |  | 23
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 |  | 0
Age, Continuous [Median (Full Range); unit: years] | 3 [2 to 7] | 17.5 [12 to 26] | 14 [3 to 22] | 14 [10 to 29] | 17 [8 to 28] | 10.5 [2 to 30] | 14.5 [4 to 26] | 14.5 [3 to 24] | 7 [4 to 14] |  | 13 [2 to 30]
Gender [Number; unit: participants]
  Female | 3 | 6 | 6 | 6 | 6 | 8 | 9 | 3 | 8 |  | 55
  Male | 7 | 6 | 15 | 4 | 8 | 12 | 1 | 7 | 1 |  | 61
Ethnicity (NIH/OMB) [Number; unit: participants]
  Hispanic or Latino | 1 | 4 | 3 | 2 | 0 | 2 | 1 | 1 | 1 |  | 15
  Not Hispanic or Latino | 7 | 8 | 17 | 8 | 14 | 18 | 8 | 9 | 7 |  | 96
  Unknown or Not Reported | 2 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 |  | 5
Race (NIH/OMB) [Number; unit: participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 |  | 0
  Asian | 1 | 1 | 1 | 0 | 1 | 0 | 1 | 0 | 0 |  | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 |  | 0
  Black or African American | 2 | 0 | 4 | 1 | 0 | 3 | 0 | 3 | 2 |  | 15
  White | 4 | 9 | 13 | 8 | 12 | 16 | 6 | 6 | 6 |  | 80
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 |  | 0
  Unknown or Not Reported | 3 | 2 | 3 | 1 | 1 | 1 | 3 | 1 | 1 |  | 16
Region of Enrollment [Number; unit: participants]
  United States | 10 | 11 | 18 | 9 | 14 | 19 | 9 | 10 | 8 |  | 108
  Canada | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 |  | 2
  Australia | 0 | 0 | 3 | 0 | 0 | 1 | 1 | 0 | 1 |  | 6

OUTCOME MEASURES:

1. Primary Outcome: Disease Response
Description: Response rates will be calculated as the percent of patients whose best response is a Complete Response (CR) or Partial Response (PR).
Time Frame: First six treatment cycles - 24 weeks
Population: Grp 2, 12 enrolled 1 ineligible, 1 progressive disease prior to first dose of therapy. Grp 3, 21 enrolled, 1 ineligible. Grp 5, 14 enrolled, 1 ineligible. Grp 8, 10 enrolled, 1 not evaluable (patient didn't receive any drug).
Measure: Number; unit: patient
Arm/Group | Group 1 - Recurrent or Refractory Hepatoblastoma | Group 2 - Recurrent or Refractory Synovial Sarcoma | Group 3 - Recurrent or Refractory Rhabdomyosarcoma | Grp 4-Recurrent or Refractory Adrenocortical Carcinoma | Grp 5-Ewing Sarcoma/Peripheral Primitive Neuroectodermal Tumor | Grp 6 - Neuroblastoma-MIBG Positive Without Measurable Disease | Grp 7-Neuroblastoma With Measurable Disease | Group 8 - Recurrent Osteosarcoma | Group 9 - Recurrent or Refractory Wilms Tumor | Group 10 - Recurrent or Refractory Retinoblastoma
Number analyzed (Participants) | 10 | 10 | 20 | 10 | 13 | 20 | 10 | 9 | 9 | 0
patient
  Non-Responder | 10 | 10 | 19 | 10 | 11 | 16 | 10 | 9 | 9 |
  Responder | 0 | 0 | 1 | 0 | 2 | 4 | 0 | 0 | 0 |

ADVERSE EVENTS:
Time Frame: Group 2, 12 enrolled 1 ineligible, 1 progressive disease prior to first dose of therapy. Group 3, 21 enrolled, 1 ineligible. Group 5, 14 enrolled, 1 ineligible. Group 8, 10 enrolled, 1 not evaluable (patient didn't receive any drug).
Description: SAE field contains NCI CTCAEs submitted via expedited reporting (NCI AdEERs / CAeRs). The AE field contains grade 3 and higher CTCAEs reported on study excluding those that were reported as SAEs.
Arm/Group | Group 1 - Recurrent or Refractory Hepatoblastoma | Group 2 - Recurrent or Refractory Synovial Sarcoma | Group 3 - Recurrent or Refractory Rhabdomyosarcoma | Grp 4-Recurrent or Refractory Adrenocortical Carcinoma | Grp 5-Ewing Sarcoma/Peripheral Primitive Neuroectodermal Tumor | Grp 6 - Neuroblastoma-MIBG Positive Without Measurable Disease | Grp 7-Neuroblastoma With Measurable Disease | Group 8 - Recurrent Osteosarcoma | Group 9 - Recurrent or Refractory Wilms Tumor | Group 10 - Recurrent or Refractory Retinoblastoma
Serious Adverse Events (participants affected / at risk) | 7/10 | 3/10 | 4/20 | 5/10 | 5/13 | 5/20 | 4/10 | 4/9 | 5/9 | 0/0
Other Adverse Events (participants affected / at risk) | 5/10 | 7/10 | 14/20 | 5/10 | 8/13 | 9/20 | 9/10 | 5/9 | 9/9 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1 - Recurrent or Refractory Hepatoblastoma (N=10) | Group 2 - Recurrent or Refractory Synovial Sarcoma (N=10) | Group 3 - Recurrent or Refractory Rhabdomyosarcoma (N=20) | Grp 4-Recurrent or Refractory Adrenocortical Carcinoma (N=10) | Grp 5-Ewing Sarcoma/Peripheral Primitive Neuroectodermal Tumor (N=13) | Grp 6 - Neuroblastoma-MIBG Positive Without Measurable Disease (N=20) | Grp 7-Neuroblastoma With Measurable Disease (N=10) | Group 8 - Recurrent Osteosarcoma (N=9) | Group 9 - Recurrent or Refractory Wilms Tumor (N=9) | Group 10 - Recurrent or Refractory Retinoblastoma (N=0)
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Acidosis (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 2 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Anaphylaxis (Immune system disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Anemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Anorexia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Appendicitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Asystole (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Bladder infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Chest wall pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Confusion (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Creatinine increased (Investigations) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cystitis noninfective (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Death NOS (General disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Device related infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Diarrhea (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dry mouth (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
GGT increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hyperkalemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hypermagnesemia (Metabolism and nutrition disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Hyperuricemia (Metabolism and nutrition disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypocalcemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hypoglycemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hypokalemia (Metabolism and nutrition disorders) | 2 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Hypophosphatemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Hypotension (Vascular disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hypothyroidism (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Infections and infestations - Other (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 2 | 0
INR increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Intra-abdominal hemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Investigations - Other (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Lymphocyte count decreased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Neutrophil count decreased (Investigations) | 2 | 1 | 1 | 1 | 1 | 0 | 1 | 1 | 1 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Pelvic pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Platelet count decreased (Investigations) | 0 | 0 | 2 | 0 | 0 | 1 | 1 | 1 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Postoperative hemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Proteinuria (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Renal and urinary disorders - Other (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Respiratory, thoracic and mediastinal disorders - Other (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Upper respiratory infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Urinary tract obstruction (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
White blood cell decreased (Investigations) | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1 - Recurrent or Refractory Hepatoblastoma (N=10) | Group 2 - Recurrent or Refractory Synovial Sarcoma (N=10) | Group 3 - Recurrent or Refractory Rhabdomyosarcoma (N=20) | Grp 4-Recurrent or Refractory Adrenocortical Carcinoma (N=10) | Grp 5-Ewing Sarcoma/Peripheral Primitive Neuroectodermal Tumor (N=13) | Grp 6 - Neuroblastoma-MIBG Positive Without Measurable Disease (N=20) | Grp 7-Neuroblastoma With Measurable Disease (N=10) | Group 8 - Recurrent Osteosarcoma (N=9) | Group 9 - Recurrent or Refractory Wilms Tumor (N=9) | Group 10 - Recurrent or Refractory Retinoblastoma (N=0)
Abdominal pain (Gastrointestinal disorders) | 1 | 1 | 0 | 1 | 0 | 1 | 1 | 0 | 1 | 0
Agitation (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 3 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Alkaline phosphatase increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Allergic reaction (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Anemia (Blood and lymphatic system disorders) | 1 | 0 | 4 | 1 | 2 | 2 | 2 | 2 | 2 | 0
Anorexia (Metabolism and nutrition disorders) | 1 | 1 | 1 | 0 | 1 | 1 | 0 | 0 | 1 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 2 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Bladder infection (Infections and infestations) | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Bladder spasm (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood bilirubin increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Bruising (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Burn (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cognitive disturbance (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Creatinine increased (Investigations) | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Cushingoid (Endocrine disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cytokine release syndrome (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0
Depression (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Diarrhea (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Duodenal obstruction (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Endocrine disorders - Other (Endocrine disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Extrapyramidal disorder (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Eye infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 1 | 2 | 0 | 4 | 2 | 1 | 0 | 1 | 0
Fever (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0
Fibrinogen decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Gait disturbance (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
GGT increased (Investigations) | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 0 | 1 | 2 | 1 | 1 | 2 | 0 | 2 | 1 | 0
Hyperkalemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hypertriglyceridemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 | 2 | 1 | 2 | 0 | 0 | 0 | 1 | 0 | 0
Hypocalcemia (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0
Hypoglycemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypomagnesemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hyponatremia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Hypophosphatemia (Metabolism and nutrition disorders) | 0 | 2 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Joint effusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Lung infection (Infections and infestations) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Lymphocyte count decreased (Investigations) | 1 | 2 | 3 | 0 | 4 | 2 | 0 | 0 | 2 | 0
Memory impairment (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Middle ear inflammation (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Mucositis oral (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Neutrophil count decreased (Investigations) | 0 | 1 | 5 | 1 | 0 | 3 | 0 | 3 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Otitis externa (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Otitis media (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pain (General disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1 | 0 | 1 | 1 | 1 | 2 | 0 | 0
Pelvic pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Peripheral motor neuropathy (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 0 | 2 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Platelet count decreased (Investigations) | 1 | 0 | 0 | 0 | 2 | 4 | 1 | 0 | 1 | 0
Proteinuria (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Psychosis (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Purpura (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Respiratory, thoracic and mediastinal disorders - Other (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Skin infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Toothache (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Tracheitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Upper respiratory infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 3 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Urinary tract pain (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 2 | 2 | 0 | 0 | 0 | 1 | 0 | 0
Weight loss (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
White blood cell decreased (Investigations) | 0 | 0 | 4 | 0 | 1 | 1 | 1 | 0 | 0 | 0
Wound infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less